CLINICAL TRIAL: NCT07067957
Title: Prevalence of Functional Lower Urinary Tract Voiding Dysfunction in School-Aged Children
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Elmaadawy, Lecturer of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1073/1/25
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Voiding Dysfunction; Urinary Incontinence; Urination Disorders; Lower Urinary Tract Symptoms; Pediatrics; Constipation
MeSH Terms: conditions — Urinary Incontinence; Urination Disorders; Lower Urinary Tract Symptoms; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: School-aged Children
  Interventions: Other: Arabic Dysfunctional Voiding Symptom Score Questionnaire (DVSS)

INTERVENTIONS:
Other: Arabic Dysfunctional Voiding Symptom Score Questionnaire (DVSS) — A validated Arabic version of the Dysfunctional Voiding Symptom Score Questionnaire (DVSS) questionnaire will be used to screen children for symptoms of lower urinary tract dysfunction. It includes 10 items assessing urinary and bowel habits.

SUMMARY:
The aim of this study is to investigate the prevalence of voiding disorders and the related risk factors for the primary school-age children in El Ghrbia Government

DETAILED DESCRIPTION:
Lower urinary tract dysfunction (LUTD) is classified as a storage and voiding symptoms. Storage symptoms are increased or decreased urinary frequency, urinary incontinence, urinary urgency, and nocturia. Voiding symptoms are classified as hesitation, straining, weak stream, and intermittency. Other symptoms are holding maneuvers, feeling of incomplete emptying, postmicturition dribble, and genital and lower urinary tract pain. Constipation and/or fecal incontinence are closely related to LUTD, among children over 5 years due to functional or nonorganic causes.

The exact prevalence of the lower urinary tract dysfunction (LUTD) is unknown, approximately 20% to 30% of children in the world have symptoms associated with voiding disorders. In epidemiological studies, this ratio is between 2.1% and 19.2% in school-age children.Due to the modern lifestyle, the prevalence increases secondary to changes in toilet training and habits.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-14 years old in our locality.

Exclusion Criteria:

* Children with known anatomical anomalies of urinary tract
* Children with known neurological anomalies (spinal dysraphism, multiple sclerosis, lumbar or spinal neuritis……… etc)
* Children with history of back or lower urinary tract trauma
* Parents who refuse participation

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: School-aged children (4-14 years) attending primary schools in El Gharbia Governorate, Egypt, during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Voiding Dysfunction | 1 Hour after completion of the questionnaire
  Prevalence of Voiding Dysfunction Among School-Aged Children will be Measured using the validated Arabic version of the Dysfunctional Voiding Symptom Score (DVSS). Children with a score above the diagnostic threshold will be considered as having voiding dysfunction.

SECONDARY OUTCOMES:
Frequency of Constipation in Children With Voiding Dysfunction | 1 Hour after completion of the questionnaire
  Constipation history will be identified through the Dysfunctional Voiding Symptom Score (DVSS) questionnaire and confirmed during clinical evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author